CLINICAL TRIAL: NCT03039153
Title: The Peripheral Nerve Blocks Analgesia in Patients Undergoing Knee Replacement Surgery is a Risk Factor for the Development of Pressure Sores at the Heel? Retrospective Cohort Study
Brief Title: Pressure Ulcers in Knee Replacement Surgery
Acronym: peripress
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 0000669
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Knee Osteoarthritis; Pressure Ulcer
MeSH Terms: conditions — Osteoarthritis, Knee; Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
From the point of view of nursing to know exactly the different risk factors for the onset of pressure ulcers is very important as it allows to accurately orient preventive care interventions.

All the variable that could influence the development of pressure ulcer in patients undergoing knee replacement surgery are identified and collected: age, sex, body max index, risk to develop Pressure Ulcer (braden score), treatment to prevent pressure ulcers (typology of the devices used, such as air mattresses with alternating or static pressure, heel drains, frequency of mobilization carried out by both the patient care), management of eventual incontinence (use of diapers, urinary catheter), type of anesthesia, type of analgesia, length of stay, the ASA physical status classification system (ASA score), comorbidity, cancer, use of devices for controlling the position of the operated limb (foam valve), the number of physical therapy sessions actually carried out.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee joint replacement
* Secondary knee joint replacement

Exclusion Criteria:

* Cancer patients
* Adult or Senior with pressure ulcer at the heel

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing knee replacement surgery following chronic joint disease
Sampling Method: Non-Probability Sample
Enrollment: 565 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

PRIMARY OUTCOMES:
Heel Pressure Sores | every day until discharge (expected average of 6 days).
  Numbers of Participants With Heel Pressure Sores of all grade Detected According to the Classification of the Scale of the National Pressure Ulcer Advisory Panel -N.P.U.A.P.

SECONDARY OUTCOMES:
Heel Pressure Sores of grade ≥2 | every day until discharge (expected average of 6 days).
  Numbers of Participants With Heel Pressure Sores of grade ≥2 Detected According to the Classification of the Scale of the National Pressure Ulcer Advisory Panel -N.P.U.A.P.
Pressure Sores in any other site | every day until discharge (expected average of 6 days).
  Numbers of Participants With Pressure Sores in any other site Detected According to the Classification of the Scale of the National Pressure Ulcer Advisory Panel -N.P.U.A.P.
Pain | up to the first 3 days post intervention
  Pain Score on the "Numeric Rating Scale (NRS)". The NRS scale had values from 0 to 10 where zero represented no pain and 10 the worst possible pain

CONTACTS AND LOCATIONS:
Overall Officials: Gianfranco Ferrarelli, RN, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No